CLINICAL TRIAL: NCT06648980
Title: Effect of a Nutritional Supplement With Phytoglycogen on Gut-brain Axis With Focus to Perceived Stress, Mood and Sleep: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of a Nutritional Supplement With Phytoglycogen on Gut-brain Axis With Focus to Perceived Stress, Mood and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mibelle AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BTS2118/24
Record Dates: First submitted 2024-09-27; First posted 2024-10-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Perceived Stress
Keywords: perceived stress; phytoglycogen; stress; sleep; mood; gut-brain axis; BDNF

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo
- Phytoglycogen (Active Comparator): Phytoglycogen
  Interventions: Dietary Supplement: Phytoglycogen

INTERVENTIONS:
Dietary Supplement: Placebo — microcrystalline cellulose; 200 mg /day; 1 capsule/day; 1 capsule daily with breakfast
  Arms: Placebo
Dietary Supplement: Phytoglycogen — Phytoglycogen; 200 mg /day; 1 capsule/day; 1 capsule daily with breakfast
  Arms: Phytoglycogen

SUMMARY:
Aim of the study is to investigate the effects of a 8-week supplementation of a phytoglycogen on perceived stress, sleep, mood and emotional wellbeing. Additionally, stress-related biomarker will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* BMI ≥ 19 and ≤ 30 kg/m²
* Subject is in good physical and mental health as established by medical history, physical examination, vital signs, results of biochemistry, haematology
* PSQ20 total score ≥33
* Capable and willing to give written informed consent

Exclusion Criteria:

* Relevant history or presence of any severe medical disorder, potentially interfering with this study (e.g. mal absorption, chronic gastro-intestinal diseases (colitis ulcerosa, Crohn's IBS, peptic ulcers, celiac disease), depression, diabetes, heavy liver disease, immunodeficiency, pancreas insufficiency, acute cancers within last 3 years except basal cell carcinoma of the skin, etc.)
* A significant CVD event within last 3 mo. incl. myocardial infarction, stroke, congestive heart failure
* Regular intake of drugs possibly interfering with this study (e.g. antidepressants, soporifics) within 3 months prior to study start or during study (stable and controlled L-Thyroxin intake would be allowed)
* Regular intake of supplements possibly interfering with this study (e.g. cannabidiol, St. John's wort, melatonin, dietary fiber supplements, probiotics etc.) within 4 weeks prior to study start or during the study (stable vitamin D intake would be allowed)
* Vegan nutrition
* Smoker > 10 cigarettes / day
* Blood donation 4 weeks prior to screening visit and during the study
* Known pregnancy, breast feeding or intention to become pregnant during the study
* Alcohol or drug abuse
* Participation in another clinical study within the last 4 weeks and concurrent participation in another clinical study
* Relevant allergy or known hypersensitivity against compounds of the study products
* Subjects considered inappropriate for the study by investigators, including subjects who are unable or unwilling to show compliance with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Impact on perceived stress (PSQ20) | 8 weeks
  * PSQ = perceived stress questionnaire;
  * higher scores indicate higher stress levels
  * the value range is 0-100

SECONDARY OUTCOMES:
Impact on perceived stress (PSQ20) | 4 weeks
  * PSQ = perceived stress questionnaire;
  * higher scores indicate higher stress levels
  * the value range is 0-100
Impact on mood (ASTS+VT) | 4 weeks
  ASTS:
  - aktuelle Stimmungsskala (ger.) = current mood scale (eng.)
  VT:
  - additional items to calculate subscales 'vigour' and 'tension'
  seven-point rating scale; value range: 19-133; higher values represent a more negative mood state
Impact on mood (ASTS+VT) | 8 weeks
  ASTS:
  - aktuelle Stimmungsskala (ger.) = current mood scale (eng.)
  VT:
  - additional items to calculate subscales 'vigour' and 'tension'
  seven-point rating scale; value range: 19-133; higher values represent a more negative mood state
Impact on sleep (Sleep Questionnaire B/R) | 8 weeks
  Sleep Questionnaire (Schlaffragebogen B/R)
  * 31 questions
  * refers to the last two weeks
  * 12 subscales
  Part B; revised Value range for subscales: 1-5 higher values represent more intense characteristics
Impact on quality of life (SF-36) | 8 weeks
  * short form 36 (SF-36) health survey
  * assessment of quality of life
  * value range is 0-100
  * higher total scores indicate a better quality of life
Global Assessment | 8 weeks
  * subjective feeling of improvement of perceived stress
  * answer options: 'yes' or 'no';
Blood biomarker | 8 weeks
  BDNF (brain derived neurotrophic factor) and hsCRP
Impact on emotions (App evaluating emotions) | 8 weeks
  * assessment of baseline emotions and triggered emotional change
  * 5 dimensions are covered

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No